CLINICAL TRIAL: NCT00728767
Title: Brief Intervention for Heavy Drinkers - a Randomized Controlled Trial
Brief Title: Brief Intervention for Heavy Drinkers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Board of Health, Denmark (Other Government)
Responsible Party: Kit Broholm, National Board of Health Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIPH - 1948
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2009-08

CONDITIONS: Alcohol Abuse
Keywords: Heavy drinking; Brief intervention; Alcohol prevention; Randomized trial; Motivational interviewing; Intervention Studies; prevention & control
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Brief intervention
- 2 (Placebo Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Brief intervention — The intervention consists of a brief conversation based on the principles of motivational interviewing, including Rollnicks scales to assess the motivation and importance for change. The intervention has duration of about 10 minutes and qualifies as a hybrid between a minimal intervention and a brief intervention.
  The intervention also consists of two leaflets ('Good advice about drinking less' and 'Learn more about alcohol') on the harmful in having an alcohol above recommended limits, and a sheet about local alcohol treatment possibilities.
  The Intervention group is also offered a brief telephone follow up call 4 weeks later. The purpose of this is to maintain the participant's motivation to reduce drinking.
  Employees had been instructed to ask these questions during the intervention: "What are you already doing to restrain your drinking?" And "What can you do more?"
  Arms: 1
Other: Control group — The intervention consists of two leaflets ('Good advice about drinking less' and 'Learn more about alcohol') on the harmful in having an alcohol use above the recommended limits, and a sheet about local alcohol treatment possibilities.
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether a brief intervention (a short conversation build on the principles of motivational interviewing) is effective in lowering self reported alcohol use in heavy drinkers.

DETAILED DESCRIPTION:
Background and purpose:

The Danish national board of Health has awarded 5.6 million DKR to two studies that will test methods that can be used for effective and early detection of heavy drinkers. The study will be carried out in 9 Danish municipalities in 2008. The study is part of the 'Diet, Smoking, Alcohol and Exercise' nationwide health study of the Danish population. It takes place in 13 municipalities in 2007 and 2008.

The study will determine whether a brief intervention is effective in lowering self reported alcohol use in heavy drinkers.

Design:

The experiment is designed as a randomized controlled trial, where heavy drinkers will be allocated to either:

A) a intervention group receiving a short (about 10 minutes) motivational conversation (build on the principles of motivational interviewing) and two leaflets about alcohol ('Good advice about drinking less' and 'Learn more about alcohol') and a sheet about local alcohol treatment possibilities. The Intervention group is also offered a brief telephone follow up call 4 weeks later. The purpose of this is to maintain the participant's motivation to reduce drinking.

B) a control group receiving two leaflets about alcohol ('Good advice about drinking less' and 'Learn more about alcohol') and a sheet about local alcohol treatment possibilities.

The study will take place in premises linked to the 'Diet, Smoking, Alcohol and Exercise' nationwide health study.

After 6 and 12 months there will be follow-up and the participants will receive a questionnaire with questions about their alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be invited to the Danish 'Diet, Smoking, Alcohol and Exercise' nationwide health study.
* Participants must have responded to an Internet questionnaire.
* Participants must have a weekly alcohol consumption above the recommended Danish limits (168 grams of alcohol for women, 252 grams of alcohol for men).

Exclusion Criteria:

* Weekly alcohol consumption less than 168 grams of alcohol for women and 252 grams of alcohol for men.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction of 25% in self reported alcohol consumption with an average volume of approximately 38-41 grams alcohol per week in the intervention group. In the control group we expect that 10% will reduce their consumption equivalent. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders B. Gottlieb Hansen, cand.techn.soc, Principal Investigator — University of Southern Denmark, National Institute of Public Health
Locations (9):
- Denmark (9):
  - The municipality of Naestved, Næstved, Næstved
  - The municipiality of Aeroe, Aeroeskoebing
  - The municipiality of Albertslund, Albertslund
  - The municipiality of Broendby, Brøndby
  - The municipiality of Frederiksberg, Frederiksberg
  - The municipality of Guldborgsund, Nykøbing Falster
  - The municipiality of Faaborg-Midtfyn, Ringe
  - The municipiality of Silkeborg, Silkeborg
  - The municipiality of Varde, Varde

REFERENCES:
- [Derived] Hansen AB, Becker U, Nielsen AS, Gronbaek M, Tolstrup JS. Brief alcohol intervention by newly trained workers versus leaflets: comparison of effect in older heavy drinkers identified in a population health examination survey: a randomized controlled trial. Alcohol Alcohol. 2012 Jan-Feb;47(1):25-32. doi: 10.1093/alcalc/agr140. Epub 2011 Sep 22. PMID 21949192